CLINICAL TRIAL: NCT00857766
Title: A Randomized, Double-Blind, Parallel-Group, 16-Week Study to Evaluate the Effect of Fluticasone Propionate/Salmeterol DISKUS® 250/50mcg BID and Placebo on Arterial Stiffness in Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: A 16-Week Study to Evaluate the Effect of Advair DISKUS™ 250/50mcg on Arterial Stiffness in Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 112355
Record Dates: First submitted 2009-03-05; First posted 2009-03-09 (Estimated); Results first posted 2010-12-23 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2016-12

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Chronic Obstructive Pulmonary Disease; arterial stiffness; Computed Tomography; pulse wave velocity; Pulse wave analysis
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- ADVAIR DISKUS (Active Comparator): Subjects receive blinded Fluticasone Propionate/Salmeterol. At 4 months subjects will receive open label SPIRIVA HANDIHALER
  Interventions: Drug: ADVAIR DISKUS™ 250/50mcg
- Placebo (Placebo Comparator): Subjects will receive placebo ADVAIR DISKUS. At 4 months subjects will receive open label SPIRIVA HANDIHALER
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: ADVAIR DISKUS™ 250/50mcg — ADVAIR DISKUS™ 250/50mcg is indicated for the twice-daily maintenance treatment of airflow obstruction in patients with chronic obstructive pulmonary disease (COPD), including chronic bronchitis and/or emphysema. ADVAIR DISKUS™ 250/50mcg is also indicated to reduce exacerbations of COPD in patients with a history of exacerbations.
  Arms: ADVAIR DISKUS
Other: Placebo — COPD subjects-Placebo DISKUS
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate in patients with Chronic Obstructive Pulmonary Disease (COPD) if Advair DISKUS™ 250/50mcg BID modifies arterial stiffness which is a measure associated with risk of heart disease.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo controlled study to evaluate the effect of Fluticasone Propionate/Salmeterol DISKUS 250/50mcg (FSC) BID on arterial stiffness in COPD subjects. Following a 1 to 14 day run-in period, approximately 250 subjects will be randomly assigned to double-blind treatment for 12 weeks. After the 12 week treatment period, subjects in both treatment arms will receive open label Tiotropium bromide Handihaler18mcg (Tio)QD for 4 weeks in addition to their continued study drug (either FSC250/50 or placebo). The primary measure of efficacy is Pulse Wave Velocity (PWV) at Endpoint. Secondary efficacy measures include Augmentation Index (AIx), Biomarkers of cardiovascular disease, measures of lung function. (e.g. FEV1). Safety will be assessed through the collection of adverse events and COPD exacerbations. Exploratory endpoints include the effect of Tiotropium on PWV and AIx when added to placebo or FSC. Treatment groups will be stratified based on current smoking status. There will be a total of 6 study visits (screening, randomization, and after 4, 8, 12 and 16 weeks of treatment). A follow-up phone contact for collection of adverse event and pregnancy information (if applicable) will be conducted approximately 14 days following the last study visit.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated written informed consent obtained from the subject and/or subject's legally acceptable representative prior to study participation.
* Males or females greater then or equal to 50 years of age.
* A post-albuterol FEV1/FVC ratio of < or equal to 0.70
* A post-albuterol FEV1 < 80% of predicted normal.
* Patients can be current or fomer smoker and must have a cigarette smoking history of > greater then or equal to 10 pack-years .

Exclusion Criteria:

* A current diagnosis of asthma
* A body mass index (BMI) of > or equal to 35kg/m2
* A respiratory diagnosis other than COPD (e.g., lung cancer, bronchiectasis, sarcoidosis, tuberculosis, lung fibrosis).

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2009-03; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (24):
- United States (24):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Jasper, Alabama
  - GSK Investigational Site, Mobile, Alabama
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Torrance, California
  - GSK Investigational Site, Hartford, Connecticut
  - GSK Investigational Site, Coeur d'Alene, Idaho
  - GSK Investigational Site, Sunset, Louisiana
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Chesterfield, Missouri
  - GSK Investigational Site, Saint Charles, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Downington, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Gaffney, South Carolina
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Union, South Carolina
  - GSK Investigational Site, Johnson City, Tennessee
  - GSK Investigational Site, Spokane, Washington
  - GSK Investigational Site, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Dransfield MT, Cockcroft JR, Townsend RR, Coxson HO, Sharma SS, Rubin DB, Emmett AH, Cicale MJ, Crater GD, Martinez FJ. Effect of fluticasone propionate/salmeterol on arterial stiffness in patients with COPD. Respir Med. 2011 Sep;105(9):1322-30. doi: 10.1016/j.rmed.2011.05.016. Epub 2011 Jun 22. PMID 21696934
- [Derived] Bhatt SP, Cole AG, Wells JM, Nath H, Watts JR, Cockcroft JR, Dransfield MT. Determinants of arterial stiffness in COPD. BMC Pulm Med. 2014 Jan 4;14:1. doi: 10.1186/1471-2466-14-1. PMID 24387157
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 112355 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 112355 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 112355 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 112355 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 112355 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 112355 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 112355 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- FSC DISKUS 250/50 mcg: Fluticasone Propionate/Salmeterol (FSC) DISKUS 250/50 micrograms (mcg) twice daily. At Visit 5 (Week 12), participants received open-label Tiotropium inhalation capsules 18 mcg per dose via Handihaler inhalation device.
- Matching Placebo: Matching placebo DISKUS twice daily. At Visit 5 (Week 12), participants received open-label Tiotropium inhalation capsules 18 mcg per dose via Handihaler inhalation device.
Period: Overall Study
Arm/Group | FSC DISKUS 250/50 mcg | Matching Placebo
Started | 123 | 126
Completed | 92 | 96
Not Completed | 31 | 30
Not completed — Adverse Event | 13 | 12
Not completed — Protocol Violation | 11 | 11
Not completed — Lost to Follow-up | 1 | 0
Not completed — Investigator Discretion | 2 | 3
Not completed — Participant Withdrew Consent | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FSC DISKUS 250/50 mcg | Matching Placebo | Total
Number analyzed (Participants) | 123 | 126 | 249
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.6 (8.92) | 63.5 (7.88) | 63.5 (8.40)
Gender [Count of Participants; unit: Participants]
  Female | 55 | 52 | 107
  Male | 68 | 74 | 142
Race/Ethnicity, Customized [Number; unit: participants]
  African American/African Heritage | 7 | 9 | 16
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 1 | 1 | 2
  White | 114 | 114 | 228

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Aortic Pulse Wave Velocity (aPWV) at the 12-Week Endpoint
Description: The 12-week Endpoint is defined as the last scheduled measurement of PWV during the 12-week double-blind treatment period (from Visits 3-5; Weeks 4, 8, and 12, respectively), and Baseline is defined as the PWV measure from Visit 2 (Randomization). Change from Baseline was calculated as the Endpoint value minus the Baseline Value. PWV is used as a measure of arterial stiffness, which is a measure of the cushioning functioning of major vessels like the aorta. The velocity of the PW along an artery is dependent on the stiffness of that artery.
Time Frame: Baseline and the 12-Week Endpoint (up to Week 12)
Population: Intent-to-Treat (ITT) Population: all participants who were randomized to study drug. The number analyzed at baseline is different from that at the 12-week endpoint due to participant withdrawal. Data are missing for some participants in the ITT Population.
Measure: Mean (Standard Error); unit: meters per second (m/s)
Arm/Group | FSC DISKUS 250/50 mcg | Matching Placebo
Number analyzed (Participants) | 118 | 122
meters per second (m/s)
  Baseline, n=118, 122 | 10.06 (0.26) | 9.87 (0.25)
  12-Week Endpoint, n=113, 110 | 9.83 (0.24) | 9.95 (0.26)
  Change from Baseline | -0.24 (0.194) | 0.13 (0.157)
Statistical Analysis 1: Comparison: FSC DISKUS 250/50 mcg vs Matching Placebo; Test type: Superiority or Other; p = 0.065, ANCOVA; Least squares (LS) mean difference = -0.42, 95% CI [-0.88 to 0.03] — LS mean difference is calculated as FSC 250/50 minus Placebo and is adjusted for treatment, investigator, sex, smoking status, age, body mass index (BMI), waist circumference, treatment by sex interaction, age by BMI interaction, and baseline value

2. Secondary Outcome: Mean Change From Baseline in Augmentation Index (AIx) at the 12-Week Endpoint
Description: AIx is a surrogate measure of peripheral (not aortic) arterial resistance and is measured by analysis of the pulse wave at the radial artery. AIx = ([delta P/Pulse Pressure] x 100); delta P is defined by a notch near the peak of the pulse wave. Change from Baseline was calculated as the Endpoint value minus the Baseline Value.
Time Frame: Baseline and the 12-Week Endpoint (up to Week 12)
Population: ITT Population. The number analyzed at baseline is different from that at the 12-week endpoint due to participant withdrawal. Data are missing for some participants in the ITT Population.
Measure: Mean (Standard Error); unit: % of total height of peak pulse pressure
Arm/Group | FSC DISKUS 250/50 mcg | Matching Placebo
Number analyzed (Participants) | 121 | 122
% of total height of peak pulse pressure
  Baseline, n=121, 122 | 27.9 (0.83) | 27.8 (0.83)
  12-Week Endpoint, n=114, 111 | 27.2 (0.82) | 27.6 (0.82)
  Change from Baseline | -0.7 (0.66) | -0.4 (0.72)
Statistical Analysis 1: Comparison: FSC DISKUS 250/50 mcg vs Matching Placebo; Test type: Superiority or Other; p = 0.469, ANCOVA; Least squares analysis = -0.6, 95% CI [-2.3 to 1.1], Standard Error of Mean 0.86

3. Secondary Outcome: Mean Change From Baseline in Forced Expiratory Volume in One Second (FEV1) at the 12-Week Endpoint
Description: FEV1 is a measure of air flow via spirometry. Change from Baseline was calculated as the Endpoint value minus the Baseline Value.
Time Frame: Baseline and the 12-Week Endpoint (up to Week 12)
Population: as for outcome 2
Measure: Mean (Standard Error); unit: milliliters
Arm/Group | FSC DISKUS 250/50 mcg | Matching Placebo
Number analyzed (Participants) | 123 | 125
milliliters
  Baseline, n=123, 125 | 1444 (53.7) | 1480 (60.1)
  12-Week Endpoint, n=105, 102 | 1588 (59.6) | 1500 (61.6)
  Change from Baseline | 136 (22.0) | -3 (30.4)
Statistical Analysis 1: Comparison: FSC DISKUS 250/50 mcg vs Matching Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Least squares analysis = 127, 95% CI [57 to 197], Standard Error of Mean 35.5

ADVERSE EVENTS:
Time Frame: 16 week observation
Arm/Group | FSC DISKUS 250/50 mcg | Matching Placebo
Serious Adverse Events (participants affected / at risk) | 8/123 | 8/126
Other Adverse Events (participants affected / at risk) | 9/123 | 7/126
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FSC DISKUS 250/50 mcg (N=123) | Matching Placebo (N=126)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Pneumonia (Infections and infestations) | 3 | 0
Bronchitis (Infections and infestations) | 1 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FSC DISKUS 250/50 mcg (N=123) | Matching Placebo (N=126)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.